CLINICAL TRIAL: NCT00176839
Title: Busulfan, Cyclophosphamide, and Melphalan Followed by Allogeneic Hematopoietic Cell Transplantation in Patients With Hematological Malignancies
Brief Title: Stem Cell Transplantation for Hematological Malignancies
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Replaced by a different study
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000LS040; MT2000-12 (Other: Blood and Marrow Transplantation Program); 0005M52481 (Other: Institutional Review Board, University of Minnesota)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2013-02-13 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Leukemia, Lymphocytic, Acute; AML; MDS
Keywords: Stem Cell transplant; retransplant; hematological malignancies
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hematologic Neoplasms | interventions — Stem Cell Transplantation; Bone Marrow Transplantation; Busulfan; Cyclophosphamide; Melphalan; Granulocyte Colony-Stimulating Factor; Filgrastim; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Patients treated with therapy plan consisting of Busulfan every 6 hours on days -7 through -4, Cyclophosphamide 60 mg/kg/day IV x 2 days, Melphalan 140 mg/m on day -1, antithymocyte globulin (ATG), G-CSF (granulocyte colony-stimulating factor) and stem cell transplantation on day 0.
  Interventions: Procedure: Stem Cell Transplant; Drug: Busulfan; Drug: Cyclophosphamide; Drug: Melphalan; Drug: G-CSF; Drug: ATG

INTERVENTIONS:
Procedure: Stem Cell Transplant — Certain cancers can be treated by giving patients stem cells that come from someone else. This is called a stem-cell transplant. As part of the transplant process, patients receive high doses of chemotherapy and/or radiation to treat their underlying disease, such as cancer. As one of its effects, this treatment also kills the healthy stem cells that are already in the marrow. The transplant provides new stem cells for the patient from a healthy donor; that replace the bone marrow and allow the blood counts to recover.
  Other Names: Bone Marrow Transplant; umbilical cord transplant; hematopoietic stem cell transplant
Drug: Busulfan — Prior to transplantation, subjects will receive BUSULFAN via the central venous line, four times a day for four days (days -7 through -4).
  Other Names: Busulfex, Myleran
Drug: Cyclophosphamide — Prior to stem cell transplantation, subjects will receive CYCLOPHOSPHAMIDE via the central venous line once a day for two days on days -3 and -2.
  Other Names: Cytoxan, Neosar
Drug: Melphalan — MELPHALAN will be given via the central venous line for one day, on day -1, prior to stem cell transplantation.
  Other Names: Alkeran
Drug: G-CSF — G-CSF is to be given daily IV beginning on day +1 until ANC 2.5 x 109/L.
  Other Names: granulocyte colony-stimulating factor, Filgrastim, Neupogen
Drug: ATG — ATG will be administered to umbilical cord blood recipients.
  Other Names: antithymocyte globulin

SUMMARY:
This protocol using busulfan, cyclophosphamide and melphalan has been designed as conditioning therapy for patients receiving stem cell transplantation for acute leukemia or myelodysplastic syndrome (MDS). The hypothesis is that this new regimen will be well tolerated and will cure the patient.

DETAILED DESCRIPTION:
Subjects will be admitted to the bone marrow transplant unit and put in isolation to reduce exposure to infectious agents.

Prior to transplantation, they will receive BUSULFAN via the central venous line, four times a day for four days, CYCLOPHOSPHAMIDE via the central venous line once a day for two days, and MELPHALAN via the central venous line for one day. Busulfan, cyclophosphamide, and melphalan are given to destroy the subject's cancer. As well, these drugs will destroy their immune system to help ensure the new stem cells take and grow after transplantation.

On the day of transplantation, umbilical cord blood from the donor will be transfused via venous line. These new cells will replace the subject's bone marrow.

After transplantation, the subjects will receive Cyclosporin A and either MMF or MTX

Isolation will be continued until adequate numbers of cells are present in the blood to fight infection. Subjects will be discharged from the hospital when medically ready. They will be expected to return for follow-up to the blood and marrow transplant clinic at specific dates as determined by physicians.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of acute lymphocytic leukemia (ALL), acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) and currently be in complete remission.
* Patients must be either:
* - <18 years of age who are at least 6 months after initial hematopoietic cell transplant (HCT),
* - 19-35 years of age and at least 18 months after initial HCT, or
* - <35 years of age and have received sufficient radiation treatment to be ineligible for total body irradiation (TBI) containing preparative therapy
* Adequate major organ function including:
* - Cardiac: ejection fraction > or = 45%
* - Renal: creatinine clearance > or = 40 mL/min
* - Hepatic: no clinical evidence of hepatic failure (e.g. coagulopathy, ascites)
* - Karnofsky performance status > or = 70% or Lansky score > or = 50%
* Women of child bearing age must be using adequate birth control and have a negative pregnancy test.
* Written informed consent.

Exclusion Criteria:

* Eligible for TBI containing preparative regimen.
* Active uncontrolled infection within one week of HCT.
* Pregnant or lactating females.

Max Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2000-06-07 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret MacMillan, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was offered to patients at the time different treatment options were being discussed in the clinic or in the hospital.
Groups:
- Treatment Arm: Patients treated with therapy plan ((Busulfan, Cyclophosphamide, Melphalan, antithymocyte globulin (ATG), G-CSF (granulocyte colony-stimulating factor) and stem cell transplantation.
Period: Overall Study
Arm/Group | Treatment Arm
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Probability of Long-term Disease-free Survival (DFS)
Description: Number of participants with long-term disease free survival after being treated with busulfan (BU), cyclophosphamide (CY) and melphalan (L-PAM) followed by HCT for hematological malignancies.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 11
participants | 3

2. Secondary Outcome: Probability of Engraftment
Description: Number of participants with engraftment after being treated with busulfan (BU), cyclophosphamide (CY) and melphalan (L-PAM) followed by HCT for hematological malignancies..
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 11
participants | 10

3. Secondary Outcome: Incidence of Acute Graft-versus-host Disease (GVHD)
Description: Number of participants with acute GVHD after being treated with busulfan (BU), cyclophosphamide (CY) and melphalan (L-PAM) followed by HCT for hematological malignancies.
Time Frame: 100 days post-transplant
Measure: Number; unit: participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 11
participants | 7

4. Secondary Outcome: Incidence Chronic Graft-versus-host Disease (GVHD)
Description: Number of participants with chronic GVHD after being treated with busulfan (BU), cyclophosphamide (CY) and melphalan (L-PAM) followed by HCT for hematological malignancies.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 11
participants | 0

5. Secondary Outcome: Incidence of Regimen-related Toxicity 100 Days Post Transplant
Description: Number of participants with regimen-related toxicity 100 days post transplant after being treated with busulfan (BU), cyclophosphamide (CY) and melphalan (L-PAM) followed by HCT for hematological malignancies.
Time Frame: 100 days post-transplant
Measure: Number; unit: participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 11
participants | 3

6. Secondary Outcome: Incidence of Relapse
Description: Number of patients with relapse after being treated with busulfan (BU), cyclophosphamide (CY) and melphalan (L-PAM) followed by HCT for hematological malignancies.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 11
participants | 2

ADVERSE EVENTS:
Time Frame: 1 year post transplant.
Arm/Group | Treatment Arm
Serious Adverse Events (participants affected / at risk) | 10/11
Other Adverse Events (participants affected / at risk) | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=11)
Fungal Infection (Infections and infestations) | 1 (1)
Pulmonary Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Graft Versus Host Disease (Immune system disorders) | 7 (7)
Graft Failure (Immune system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes